CLINICAL TRIAL: NCT00699374
Title: A Multinational, Randomized, Open-Label, Phase 3 Study Of Sunitinib Malate Versus Sorafenib In Patients With Advanced Hepatocellular Carcinoma
Brief Title: Study Of Sunitinib Malate Versus Sorafenib In Patients With Inoperable Liver Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A6181170
Record Dates: First submitted 2008-06-16; First posted 2008-06-18 (Estimated); Results first posted 2013-01-14 (Estimated); Last update posted 2013-01-14 (Estimated); Status verified 2012-12

CONDITIONS: Carcinoma, Hepatocellular
Keywords: sunitinib; phase 3; randomized; hepatocellular; liver
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sunitinib; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Experimental): sunitinib arm
  Interventions: Drug: sunitinib malate
- Arm B (Active Comparator): sorafenib arm
  Interventions: Drug: sorafenib

INTERVENTIONS:
Drug: sunitinib malate — sunitinib capsules at starting dose of 37.5 mg PO daily, until disease progression, occurrence of unacceptable toxicity, or other withdrawal criteria are met. Sunitinib dosing interruptions and/or reductions are allowed based on patient tolerability.
  Other Names: Sutent®
  Arms: Arm A
Drug: sorafenib — sorafenib tablets at starting dose of 400 mg PO twice daily, until disease progression, occurrence of unacceptable toxicity, or other withdrawal criteria are met. Sorafenib dosing interruptions and/or reductions are allowed based on patient tolerability.
  Other Names: Nexavar®
  Arms: Arm B

SUMMARY:
The study will evaluate the efficacy and safety of sunitinib (Arm A), given at 37.5 mg orally once daily, compared to sorafenib (Arm B), given orally at 400 mg twice daily, in patients with inoperable liver cancer. A total number of 1200 patients will be enrolled, 600 on Arm A and 600 on Arm B. Study treatment may be adjusted based on patient tolerance. and will be given until disease progression, occurrence of unacceptable toxicity, or other withdrawal criteria are met. After discontinuation of study treatment, patients will be followed up in order to collect information on further antineoplastic therapy and survival.

DETAILED DESCRIPTION:
This study was terminated on April 22th, 2010, based on a higher incidence of serious adverse events in the sunitinib arm compared to the sorafenib arm, and the fact that sunitinib did not meet the criteria to demonstrate that it was either superior or non-inferior to sorafenib in the survival of patients with advanced hepatocellular cancer. Patients on sunitinib who are judged by the investigator as receiving clinical benefit may chose to remain on study and continue treatment with sunitinib until clinical benefit as per the investigator's judgment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed diagnosis of hepatocellular carcinoma
* presence of measurable disease by radiographic imaging
* Child-Pugh class A
* ECOG PS 0 or 1
* adequate organ function.

Exclusion Criteria:

* Prior treatment with any systemic treatment for hepatocellular carcinoma
* prior local treatment within 4 weeks from entry
* presence of clinically relevant ascites
* severe hemorrhage <4 weeks of starting study treatment
* known HIV or serious acute or chronic illness
* current treatment on another clinical trial
* pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1075 (Actual)
Dates: Start 2008-07; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (139):
- United States (25):
  - Pfizer Investigational Site, Fountain Valley, California
  - Pfizer Investigational Site, La Jolla, California
  - Pfizer Investigational Site, Orange, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Ringgold, Georgia
  - Pfizer Investigational Site, Iowa City, Iowa
  - Pfizer Investigational Site, Crestview Hills, Kentucky
  - Pfizer Investigational Site, The Bronx, New York
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Fairfield, Ohio
  - Pfizer Investigational Site, Hamilton, Ohio
  - Pfizer Investigational Site, Chattanooga, Tennessee
  - Pfizer Investigational Site, Franklin, Tennessee
  - Pfizer Investigational Site, Gallatin, Tennessee
  - Pfizer Investigational Site, Hermitage, Tennessee
  - Pfizer Investigational Site, Hixson, Tennessee
  - Pfizer Investigational Site, Lebanon, Tennessee
  - Pfizer Investigational Site, Murfreesboro, Tennessee
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, Smyrna, Tennessee
  - Pfizer Investigational Site, Mechanicsville, Virginia
  - Pfizer Investigational Site, Midlothian, Virginia
  - Pfizer Investigational Site, Richmond, Virginia
  - Pfizer Investigational Site, Seattle, Washington
- Australia (5):
  - Pfizer Investigational Site, Concord, New South Wales
  - Pfizer Investigational Site, Elizabeth Vale, South Australia
  - Pfizer Investigational Site, Woodville South, South Australia
  - Pfizer Investigational Site, Melbourne, Victoria
  - Pfizer Investigational Site, Parkville, Victoria
- Belgium (2):
  - Pfizer Investigational Site, Brussels
  - Pfizer Investigational Site, Ghent
- Canada (5):
  - Pfizer Investigational Site, Calgary, Alberta
  - Pfizer Investigational Site, Vancouver, British Columbia
  - Pfizer Investigational Site, Kingston, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Montreal, Quebec
- China (13):
  - Pfizer Investigational Site, Hefei, Anhui
  - Pfizer Investigational Site, Fuzhou, Fujian
  - Pfizer Investigational Site, Guangzhou, Guangdong
  - Pfizer Investigational Site, Nanning, Guangxi
  - Pfizer Investigational Site, Wuhan, Hubei
  - Pfizer Investigational Site, Nanjing, Jiangsu
  - Pfizer Investigational Site, Chengdu, Sichuan
  - Pfizer Investigational Site, Hangzhou, Zhejiang
  - Pfizer Investigational Site, Beijing
  - Pfizer Investigational Site, Chongqing
  - Pfizer Investigational Site, Guangzhou
  - Pfizer Investigational Site, Nanjing
  - Pfizer Investigational Site, Shanghai
- France (12):
  - Pfizer Investigational Site, Amiens
  - Pfizer Investigational Site, Bordeaux
  - Pfizer Investigational Site, Clichy
  - Pfizer Investigational Site, Créteil
  - Pfizer Investigational Site, Lille
  - Pfizer Investigational Site, Nice
  - Pfizer Investigational Site, Paris
  - Pfizer Investigational Site, Saint-Herblain
  - Pfizer Investigational Site, Strasbourg
  - Pfizer Investigational Site, Toulouse
  - Pfizer Investigational Site, Vandœuvre-lès-Nancy
  - Pfizer Investigational Site, Villejuif
- Germany (4):
  - Pfizer Investigational Site, Hamburg
  - Pfizer Investigational Site, Hanover
  - Pfizer Investigational Site, Mainz
  - Pfizer Investigational Site, München
- Hong Kong (4):
  - Pfizer Investigational Site, Tuen Mun, New Territories, Hong Kong
  - Pfizer Investigational Site, Hong Hong
  - Pfizer Investigational Site, Kowloon
  - Pfizer Investigational Site, Shatin, New Territories
- Italy (9):
  - Pfizer Investigational Site, Meldola, FC
  - Pfizer Investigational Site, Bari
  - Pfizer Investigational Site, Bologna
  - Pfizer Investigational Site, Cattolica (RN)
  - Pfizer Investigational Site, Milan
  - Pfizer Investigational Site, Padua
  - Pfizer Investigational Site, Pavia
  - Pfizer Investigational Site, Ravenna
  - Pfizer Investigational Site, Rimini
- Japan (19):
  - Pfizer Investigational Site, Nagoya, Aichi-ken
  - Pfizer Investigational Site, Chiba, Chiba
  - Pfizer Investigational Site, Kashiwa-shi, Chiba
  - Pfizer Investigational Site, Kurume, Fukuoka
  - Pfizer Investigational Site, Gifu, Gifu
  - Pfizer Investigational Site, Sapporo, Hokkaido
  - Pfizer Investigational Site, Nishinomiya, Hyōgo
  - Pfizer Investigational Site, Kanazawa, Ishikawa-ken
  - Pfizer Investigational Site, Omura-shi, Nagasaki
  - Pfizer Investigational Site, Okayama, Okayama-ken
  - Pfizer Investigational Site, Osaka, Osaka
  - Pfizer Investigational Site, Ōsaka-sayama, Osaka
  - Pfizer Investigational Site, Izunokuni-shi, Shizuoka
  - Pfizer Investigational Site, Bunkyo-ku, Tokyo
  - Pfizer Investigational Site, Chiyoda-ku, Tokyo
  - Pfizer Investigational Site, Chuo-ku, Tokyo
  - Pfizer Investigational Site, Itabashi-ku, Tokyo
  - Pfizer Investigational Site, Mitaka-shi, Tokyo
  - Pfizer Investigational Site, Setagaya-ku, Tokyo
- Malaysia (3):
  - Pfizer Investigational Site, Lembah Pantai, Kuala Lumpur
  - Pfizer Investigational Site, Subang Jaya, Selangor
  - Pfizer Investigational Site, Kuala Lumpur
- Philippines (5):
  - Pfizer Investigational Site, Cebu City, Cebu
  - Pfizer Investigational Site, Cebu City
  - Pfizer Investigational Site, Davao City
  - Pfizer Investigational Site, Manila
  - Pfizer Investigational Site, Quezon City
- Pfizer Investigational Site, Warsaw, Poland
- Russia (3):
  - Pfizer Investigational Site, Chelyabinsk
  - Pfizer Investigational Site, Pyatigorsk
  - Pfizer Investigational Site, Saint Petersburg
- Pfizer Investigational Site, Singapore, Singapore, Singapore
- Pfizer Investigational Site, Parktown, South Africa
- South Korea (7):
  - Pfizer Investigational Site, Goyang-si, Gyeonggi-do
  - Pfizer Investigational Site, Jeonju, Jeollabuk-do
  - Pfizer Investigational Site, Hwasun-gun, Jeollanam-do
  - Pfizer Investigational Site, Busan
  - Pfizer Investigational Site, Daegu
  - Pfizer Investigational Site, Incheon
  - Pfizer Investigational Site, Seoul
- Spain (5):
  - Pfizer Investigational Site, Palma de Mallorca, Balearic Islands
  - Pfizer Investigational Site, Sabadell, Barcelona
  - Pfizer Investigational Site, Santander, Cantabria
  - Pfizer Investigational Site, El Palmar, Murcia
  - Pfizer Investigational Site, Seville, Sevilla
- Pfizer Investigational Site, Linköping, Sweden
- Taiwan (7):
  - Pfizer Investigational Site, Pu-Tz City, Chai-Yi
  - Pfizer Investigational Site, Kwei-Shan, Taoyuan
  - Pfizer Investigational Site, Changhua
  - Pfizer Investigational Site, Kaohsiung City
  - Pfizer Investigational Site, Taichung
  - Pfizer Investigational Site, Tainan
  - Pfizer Investigational Site, Taipei
- Thailand (3):
  - Pfizer Investigational Site, Bangkok Noi, Bangkok
  - Pfizer Investigational Site, Ptumwan, Bangkok
  - Pfizer Investigational Site, Amphoe Mueang, Chiang Mai
- Turkey (Türkiye) (2):
  - Pfizer Investigational Site, Ankara
  - Pfizer Investigational Site, Istanbul
- United Kingdom (2):
  - Pfizer Investigational Site, Cambridge, Cambridgeshire
  - Pfizer Investigational Site, London

REFERENCES:
- [Derived] Abuhelwa AY, Badaoui S, Yuen HY, McKinnon RA, Ruanglertboon W, Shankaran K, Tuteja A, Sorich MJ, Hopkins AM. A clinical scoring tool validated with machine learning for predicting severe hand-foot syndrome from sorafenib in hepatocellular carcinoma. Cancer Chemother Pharmacol. 2022 Apr;89(4):479-485. doi: 10.1007/s00280-022-04411-9. Epub 2022 Feb 28. PMID 35226112
- [Derived] Cheng AL, Kang YK, Lin DY, Park JW, Kudo M, Qin S, Chung HC, Song X, Xu J, Poggi G, Omata M, Pitman Lowenthal S, Lanzalone S, Yang L, Lechuga MJ, Raymond E. Sunitinib versus sorafenib in advanced hepatocellular cancer: results of a randomized phase III trial. J Clin Oncol. 2013 Nov 10;31(32):4067-75. doi: 10.1200/JCO.2012.45.8372. Epub 2013 Sep 30. PMID 24081937
- [Derived] Koeberle D, Montemurro M, Samaras P, Majno P, Simcock M, Limacher A, Lerch S, Kovacs K, Inauen R, Hess V, Saletti P, Borner M, Roth A, Bodoky G. Continuous Sunitinib treatment in patients with advanced hepatocellular carcinoma: a Swiss Group for Clinical Cancer Research (SAKK) and Swiss Association for the Study of the Liver (SASL) multicenter phase II trial (SAKK 77/06). Oncologist. 2010;15(3):285-92. doi: 10.1634/theoncologist.2009-0316. Epub 2010 Mar 4. PMID 20203173
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6181170&StudyName=Study%20Of%20Sunitinib%20Malate%20Versus%20Sorafenib%20In%20Patients%20With%20Inoperable%20Liver%20Cancer

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant was randomized twice, once to the sorafenib arm and discontinued prior to receiving treatment and a second randomization to the sunitinib arm and dispensed treatment.
Groups:
- Sunitinib: Participants received sunitinib 37.5 milligram (mg) capsules by mouth once daily on a continuous daily dosing schedule. Dose reductions to either 25 mg or 12.5 mg were allowed. Treatment continued until disease progression, death, unacceptable toxicity, withdrawal of participant consent, need for different cancer treatment, or another withdrawal criterion was met.
- Sorafenib: Participants received sorafenib 400 mg tablets by mouth, twice daily (BID). Dose reduction to 400 mg once daily (QD) was allowed. Treatment continued until disease progression, death, unacceptable toxicity, withdrawal of participant consent, need for different cancer treatment, or another withdrawal criterion was met.
Period: Overall Study
Arm/Group | Sunitinib | Sorafenib
Started | 530 | 544
Treated | 526 | 542
Completed | 0 | 0
Not Completed | 530 | 544
Not completed — Death | 93 | 83
Not completed — Adverse Event | 70 | 67
Not completed — Global deterioration of health status | 7 | 8
Not completed — Lost to Follow-up | 3 | 5
Not completed — Withdrawal by Subject | 34 | 44
Not completed — Objective progression or relapse | 281 | 277
Not completed — Other | 18 | 15
Not completed — Protocol Violation | 2 | 6
Not completed — Study terminated by sponsor | 13 | 28
Not completed — Randomized but not treated | 4 | 2
Not completed — Died 28 days after last dose | 5 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sunitinib | Sorafenib | Total
Number analyzed (Participants) | 530 | 544 | 1074
Age Continuous [Mean (Standard Deviation); unit: Years] | 58.1 (12.86) | 58.5 (12.93) | 58.3 (12.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94 | 85 | 179
  Male | 436 | 459 | 895

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Overall survival is the duration from randomization to death. For participants who are alive, overall survival was censored at the last contact.
Time Frame: Baseline, every 4 weeks during treatment, every 8 weeks posttreatment up to Week 150
Population: Full Analysis Population, all randomized participants where participants were classifed according to the randomized treatment arm regardless of what treatment, if any, was received.
Measure: Median (95% Confidence Interval); unit: Weeks
Units Other Than Participants: Events
Arm/Group | Sunitinib | Sorafenib
Number analyzed (Participants) | 530 | 544
Number analyzed (Events) | 431 | 388
Weeks | 34.3 [31.9 to 39.9] | 43.9 [38.1 to 48.7]
Statistical Analysis 1: Comparison: Sunitinib vs Sorafenib; Test type: Superiority or Other; p = 0.9993, Log Rank — One-sided p-value based on stratified log-rank test controlling the effects of geographic region, prior transarterial chemoembolization (TACE) and tumor invasion condition; Hazard Ratio (HR) = 1.31, 95% CI 2-sided [1.14 to 1.50]

2. Secondary Outcome: Progression-Free Survival (PFS)
Description: The period from randomization until disease progression or death.
Time Frame: Baseline, every 4 weeks during treatment, every 8 weeks posttreatment up to Week 150
Population: Full Analysis Population
Measure: Median (95% Confidence Interval); unit: Weeks
Units Other Than Participants: Events
Arm/Group | Sunitinib | Sorafenib
Number analyzed (Participants) | 530 | 544
Number analyzed (Events) | 408 | 433
Weeks | 15.3 [12.1 to 17.7] | 12.6 [12.1 to 17.3]
Statistical Analysis 1: Comparison: Sunitinib vs Sorafenib; Test type: Superiority or Other; p = 0.8857, Log Rank — One-sided p-value based on stratified log-rank test controlling the effects of geographic region, prior TACE, and tumor invasion condition; Hazard Ratio (HR) = 1.13, 95% CI 2-sided [0.99 to 1.30]

3. Secondary Outcome: Time to Tumor Progression (TTP)
Description: Time in weeks from randomization to first documentation of objective tumor progression or death due to cancer, whichever comes first. Tumor progression was determined from oncologic assessment data (where data meet the criteria for progressive disease [PD])
Time Frame: Baseline, every 4 weeks during treatment, every 8 weeks posttreatment up to Week 150
Population: Full Analysis Population
Measure: Median (95% Confidence Interval); unit: Weeks
Units Other Than Participants: Events
Arm/Group | Sunitinib | Sorafenib
Number analyzed (Participants) | 530 | 544
Number analyzed (Events) | 365 | 393
Weeks | 17.7 [13.6 to 18.0] | 15.4 [12.3 to 18.1]
Statistical Analysis 1: Comparison: Sunitinib vs Sorafenib; Test type: Superiority or Other; p = 0.8459, Log Rank — One-sided p-value based on stratified log-rank test controlling the effects of geographic region, prior TACE and tumor invasion condition; Hazard Ratio (HR) = 1.13, 95% CI 2-sided [0.98 to 1.31]

4. Secondary Outcome: European Quality of Life (EQ-5D)- Health State Profile Utility Score
Description: EQ-5D: participant rated questionnaire to assess health-related quality of life in terms of a single utility score. Health State Profile component assesses level of current health for 5 domains: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression; 1 indicates better health state (no problems); 3 indicates worst health state (eg, "confined to bed"). Scoring formula assigns a utility value for each domain in the profile. Score is transformed and results in a score range -0.594 to 1.000; higher score indicates better health state.
Time Frame: Day 1 of each cycle
Population: Data were not collected per Amendment 2 to the protocol removing collection for this endpoint.
Arm/Group | Sunitinib | Sorafenib
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an adverse event (AE) and a serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Sunitinib | Sorafenib
Serious Adverse Events (participants affected / at risk) | 240/526 | 204/542
Other Adverse Events (participants affected / at risk) | 515/526 | 531/542
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib (N=526) | Sorafenib (N=542)
Anaemia (Blood and lymphatic system disorders) | 10 | 5
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 0
Splenic infarction (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 12 | 1
Angina pectoris (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 2
Bradycardia (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 2
Myocardial infarction (Cardiac disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0
Cataract (Eye disorders) | 0 | 1
Diabetic retinopathy (Eye disorders) | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 6 | 5
Abdominal pain upper (Gastrointestinal disorders) | 2 | 5
Ascites (Gastrointestinal disorders) | 12 | 6
Cheilitis (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 10 | 9
Duodenal ulcer (Gastrointestinal disorders) | 1 | 2
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 2 | 0
Faeces discoloured (Gastrointestinal disorders) | 1 | 0
Gastric antral vascular ectasia (Gastrointestinal disorders) | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 2 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 1
Gastric varices haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastritis erosive (Gastrointestinal disorders) | 1 | 0
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 12 | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 3 | 0
Glossitis (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 2 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 2
Ileus (Gastrointestinal disorders) | 2 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 1 | 2
Mesenteric vein thrombosis (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 4 | 2
Oesophageal rupture (Gastrointestinal disorders) | 1 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 1 | 0
Oesophageal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 3 | 2
Pancreatic enzyme abnormality (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 2 | 1
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 0
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 11 | 7
Vomiting (Gastrointestinal disorders) | 9 | 4
Asthenia (General disorders) | 10 | 3
Chest pain (General disorders) | 1 | 1
Condition aggravated (General disorders) | 9 | 6
Death (General disorders) | 0 | 1
Device failure (General disorders) | 1 | 0
Disease progression (General disorders) | 55 | 62
Fatigue (General disorders) | 5 | 4
General physical health deterioration (General disorders) | 3 | 6
Generalised oedema (General disorders) | 1 | 0
Hyperthermia (General disorders) | 1 | 0
Malaise (General disorders) | 2 | 0
Multi-organ failure (General disorders) | 1 | 1
Oedema peripheral (General disorders) | 1 | 0
Pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 15 | 9
Acute hepatic failure (Hepatobiliary disorders) | 1 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 2
Bile duct stone (Hepatobiliary disorders) | 0 | 1
Biliary colic (Hepatobiliary disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 1
Cholangitis acute (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 1
Hepatic failure (Hepatobiliary disorders) | 3 | 5
Hepatic function abnormal (Hepatobiliary disorders) | 4 | 4
Hepatic haemorrhage (Hepatobiliary disorders) | 1 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 1
Hepatorenal syndrome (Hepatobiliary disorders) | 0 | 2
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 3 | 2
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 1
Anaphylactic shock (Immune system disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1
Abdominal infection (Infections and infestations) | 0 | 1
Anal abscess (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 2 | 0
Biliary sepsis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Bronchopneumonia (Infections and infestations) | 0 | 1
Campylobacter infection (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 2 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Escherichia sepsis (Infections and infestations) | 1 | 0
Fungal oesophagitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 2 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 1
Hepatitis B (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1
Herpes zoster ophthalmic (Infections and infestations) | 0 | 1
Infected skin ulcer (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 1 | 1
Infectious peritonitis (Infections and infestations) | 1 | 0
Liver abscess (Infections and infestations) | 1 | 3
Lung infection (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 1 | 0
Perineal abscess (Infections and infestations) | 0 | 1
Peritonitis bacterial (Infections and infestations) | 2 | 1
Pneumonia (Infections and infestations) | 4 | 5
Pulmonary tuberculosis (Infections and infestations) | 0 | 1
Rash pustular (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1
Scrotal abscess (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 6 | 7
Septic shock (Infections and infestations) | 3 | 0
Tuberculosis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 2 | 1
Veillonella infection (Infections and infestations) | 0 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Cystitis radiation (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Traumatic liver injury (Injury, poisoning and procedural complications) | 0 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 2
Blood bilirubin increased (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 1
Liver function test abnormal (Investigations) | 0 | 2
Neutrophil count decreased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 4 | 1
White blood cell count decreased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 8 | 4
Dehydration (Metabolism and nutrition disorders) | 8 | 3
Hyperammonaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 3 | 4
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 0
Hypophagia (Metabolism and nutrition disorders) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Liver carcinoma ruptured (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Nervous system neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pharyngeal cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Tumour rupture (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Altered state of consciousness (Nervous system disorders) | 0 | 1
Cerebral artery embolism (Nervous system disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 2 | 2
Cerebral infarction (Nervous system disorders) | 2 | 0
Coma (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0
Diabetic hyperglycaemic coma (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 15 | 4
Hypoaesthesia (Nervous system disorders) | 1 | 0
Hypoglycaemic coma (Nervous system disorders) | 1 | 1
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 | 1
Lacunar infarction (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0
Paralysis (Nervous system disorders) | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 2 | 1
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 | 0
Alcoholism (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 1
Suicide attempt (Psychiatric disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Nephrotic syndrome (Renal and urinary disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 4 | 1
Renal failure acute (Renal and urinary disorders) | 2 | 1
Renal impairment (Renal and urinary disorders) | 2 | 0
Renal tubular necrosis (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0
Scrotal erythema (Reproductive system and breast disorders) | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Neuropathic ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 6 | 3
Rash (Skin and subcutaneous tissue disorders) | 0 | 2
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 2
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 | 1
Bleeding varicose vein (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Haemorrhage (Vascular disorders) | 1 | 2
Hypertension (Vascular disorders) | 1 | 0
Hypertensive crisis (Vascular disorders) | 1 | 0
Inferior vena caval occlusion (Vascular disorders) | 1 | 0
Intra-abdominal haemorrhage (Vascular disorders) | 1 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 0
Phlebitis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib (N=526) | Sorafenib (N=542)
Anaemia (Blood and lymphatic system disorders) | 79 | 47
Leukopenia (Blood and lymphatic system disorders) | 96 | 37
Neutropenia (Blood and lymphatic system disorders) | 119 | 19
Thrombocytopenia (Blood and lymphatic system disorders) | 170 | 69
Hypothyroidism (Endocrine disorders) | 30 | 7
Abdominal distension (Gastrointestinal disorders) | 90 | 56
Abdominal pain (Gastrointestinal disorders) | 121 | 105
Abdominal pain upper (Gastrointestinal disorders) | 74 | 78
Ascites (Gastrointestinal disorders) | 76 | 64
Constipation (Gastrointestinal disorders) | 90 | 81
Diarrhoea (Gastrointestinal disorders) | 248 | 254
Dyspepsia (Gastrointestinal disorders) | 53 | 39
Mouth ulceration (Gastrointestinal disorders) | 28 | 18
Nausea (Gastrointestinal disorders) | 129 | 93
Stomatitis (Gastrointestinal disorders) | 87 | 53
Vomiting (Gastrointestinal disorders) | 103 | 61
Asthenia (General disorders) | 78 | 60
Chest pain (General disorders) | 21 | 30
Face oedema (General disorders) | 35 | 5
Fatigue (General disorders) | 171 | 115
Mucosal inflammation (General disorders) | 65 | 39
Oedema (General disorders) | 46 | 23
Oedema peripheral (General disorders) | 71 | 46
Pain (General disorders) | 25 | 29
Pyrexia (General disorders) | 105 | 101
Hyperbilirubinaemia (Hepatobiliary disorders) | 59 | 43
Alanine aminotransferase increased (Investigations) | 60 | 70
Aspartate aminotransferase increased (Investigations) | 84 | 92
Blood bilirubin increased (Investigations) | 30 | 30
Gamma-glutamyltransferase increased (Investigations) | 17 | 28
Neutrophil count decreased (Investigations) | 50 | 4
Platelet count (Investigations) | 29 | 9
Platelet count decreased (Investigations) | 65 | 16
Weight decreased (Investigations) | 44 | 115
White blood cell count decreased (Investigations) | 45 | 5
Decreased appetite (Metabolism and nutrition disorders) | 233 | 187
Hypoalbuminaemia (Metabolism and nutrition disorders) | 47 | 42
Back pain (Musculoskeletal and connective tissue disorders) | 46 | 40
Pain in extremity (Musculoskeletal and connective tissue disorders) | 14 | 27
Dizziness (Nervous system disorders) | 48 | 17
Dysgeusia (Nervous system disorders) | 69 | 15
Headache (Nervous system disorders) | 43 | 40
Insomnia (Psychiatric disorders) | 60 | 54
Proteinuria (Renal and urinary disorders) | 44 | 38
Cough (Respiratory, thoracic and mediastinal disorders) | 77 | 62
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 10 | 49
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 53 | 32
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 63 | 25
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 30 | 19
Alopecia (Skin and subcutaneous tissue disorders) | 19 | 154
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 232 | 330
Pruritus (Skin and subcutaneous tissue disorders) | 34 | 58
Rash (Skin and subcutaneous tissue disorders) | 108 | 147
Yellow skin (Skin and subcutaneous tissue disorders) | 37 | 0
Hypertension (Vascular disorders) | 109 | 95

LIMITATIONS AND CAVEATS:
Study terminated early due to futility. Subsequently, EQ-5D data were not collected or analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.